CLINICAL TRIAL: NCT07300787
Title: Role of miRNA-155 and miRNA-204 in Pediatric Gastritis
Brief Title: miRNA in Pediatric Gastritis
Acronym: microRNA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Nashwa farouk Mohamed, lecturer of pediatrics, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MD 5-10-2023
Record Dates: First submitted 2025-12-07; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: miRNA-155; miRNA-204; gastritis; H.pylori
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Intervention Model Description: Gastric and duodenal biopsies specimens will obtained from patients undergoing upper gastrointestinal endoscopy for the investigation of recurrent abdominal pain. None of the patients had received any medication which may have affected gastric acidity before endoscopy. Upper GIT endoscopy was performed H.pylori was identified by Giemsa staining. Grossendoscopic findings such as peptic ulcer and erosion in the distal esophagus and stomach were regarded as pathological.Gene expression was done by quantitative reverse transcription-polymerase chain reaction (qRT-PCR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastritis group (Active Comparator): All included patients were subjected to full history taking including age, sex, residence, present illness; onset, course and duration, abdominal pain, other associated symptoms and family history. Assessment of anthropometric measurement Patients' height and weight for age and BMI percentiles were checked according to Egyptian growth curves .
  Abdominal Ultrasonography upper GIT ENDOSCOPY miRNA gene expression
  Interventions: Diagnostic Test: miRNA gene expression
- Control healthy group (Placebo Comparator): miRNA gene expression
  Interventions: Diagnostic Test: miRNA gene expression

INTERVENTIONS:
Diagnostic Test: miRNA gene expression — Gene expression was done by quantitative reverse transcription-polymerase chain reaction (qRT-PCR).
  Paraffin-embedded biopsies were sectioned into 10-μm-thick slices, two of which were deposited into 1.5-ml microcentrifuge tubes and dewaxed via immersion in xylene at 50 °C, followed by absolute and 96% ethanol.
  Extraction of total RNA (including miRNA) was performed using the Qiagen RNeasyPlus Universal Mini Kit (Qiagen, Hilden, Germany) according to manufacturer's protocol. Briefly, the samples were homogenized in QIAzol Lysis Reagent using TissueRuptor. RNA was further precipitated with chloroform, mixed with 1.5 volumes of 100% of Ethanol and following precipitation and washing steps eluted in RNase-free water. The concentration of extracted RNA was assessed using UV-spectrophotometry. MiRNA expression was quantitatively evaluated using either the TaqMan miRNA assay (Applied Biosystems, CA, USA) or SYBR Green (RNU6b) method. Approximately 20 ng of total RNA were reverse tran

SUMMARY:
The goal of this clinical trial is to assess the differential expression of miR-155 and miRNA-204 in relation to gastritis, and assess their relation with the presence of H. pylori in children.

DETAILED DESCRIPTION:
patients will be subjected to full history taking including age, sex, residence, present illness; onset, course and duration, abdominal pain, other associated symptoms and family history. Assessment of anthropometric measurement Patients' height and weight for age and BMI percentiles were checked according to Egyptian growth curves (9).

Abdominal Ultrasonography upper GITendoscopy mi RNAGene expression was done by quantitative reverse transcription-polymerase chain reaction (qRT-PCR).

ELIGIBILITY:
Inclusion Criteria:

recurrent abdominal pain warranting upper gastrointestinal endoscopy or gastroscopy including

* peptic-like dyspepsia (identified by two or more symptoms such as periodic pain, pain relief with food or antacid, pre-meal or hunger-induced pain, nausea/vomiting, and nighttime pain),
* dysmotility-like dyspepsia (characterized by abdominal distension, anorexia, weight loss, pain worsening with food/milk, and belching),
* and reflux-like dyspepsia (manifesting as heartburn, chest pain

exclusion criteria:

-patients with gastrointestinal disorders explaining abdominal pain (e.g., inflammatory bowel disease, celiac disease, functional abdominal pain)

, -patients on proton pump inhibitors, as well as those with significant medical comorbidities.

Exclusion Criteria:

-

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
differential expression of mRNA-204 and mRNA-155 in relation to gastritis, and assess their relation with the presence of H. pylori in children | in 1 month
  Gene expression was done by quantitative reverse transcription-polymerase chain reaction (qRT-PCR).
  Paraffin-embedded biopsies were sectioned into 10-μm-thick slices, two of which were deposited into 1.5-ml microcentrifuge tubes and dewaxed via immersion in xylene at 50 °C, followed by absolute and 96% ethanol.
  Extraction of total RNA (including miRNA) was performed using the Qiagen RNeasyPlus Universal Mini Kit (Qiagen, Hilden, Germany) according to manufacturer's protocol. Briefly, the samples were homogenized in QIAzol Lysis Reagent using Tissue Ruptor. RNA was further precipitated with chloroform, mixed with 1.5 volumes of 100% of Ethanol and following precipitation and washing steps eluted in RNase-free water. The concentration of extracted RNA was assessed using UV-spectrophotometry. MiRNA expression was quantitatively evaluated using either the TaqMan miRNA assay (Applied Biosystems, CA, USA) or SYBR Green (RNU6b) method.

OTHER OUTCOMES:
weight and height will be combined to report BMI in kg/m | 1 month
  Body Mass Index (BMI) is a screening tool using your weight and height to estimate body fat, calculated by dividing weight (kg) by height (m²) to categorize enrolled children into underweight, healthy, overweight, or obese, kilogram/meters^2

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bordin DS, Livzan MA, Mozgovoi SI, Gaus OV. Autoimmune Gastritis and Helicobacter pylori Infection: Molecular Mechanisms of Relationship. Int J Mol Sci. 2025 Aug 11;26(16):7737. doi: 10.3390/ijms26167737. PMID 40869058